CLINICAL TRIAL: NCT05543200
Title: A Global Registry of Treatments and Outcomes for Benign Prostatic Hyperplasia
Brief Title: BPH Global Registry
Status: Recruiting | Type: Observational
Sponsor: Société Internationale d'Urologie (Other)
Responsible Party: Sponsor
Other Study IDs: uCARE-2022-001
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: BPH, Registry, LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- All Participants: All men who have a primary diagnosis of BPH with LUTS that are prescribed BPH medications or a surgical intervention.

SUMMARY:
Benign prostatic hyperplasia (BPH) is one of the most common performed surgical procedures in urology. Over the past few decades there have been an increasing development of newer surgical treatment options. Additionally, the outcome parameters for BPH treatments have been standardized. While data are available for the initial pivotal studies, post-market release data are lacking. Under the umbrella of uCARE, we have started a prospective, ongoing international registry for recording demographics and outcomes for patients undergoing surgical treatments for BPH.

DETAILED DESCRIPTION:
Due to a growing and aging population, cases of benign prostatic hyperplasia (BPH) have been on a steady rise. Studies show that by age 80, 90% of men experience BPH. (Garraway, Lee, Collins, 1991) Thus, treatment of BPH is one of the most performed surgical procedures in urology. Over the past few decades there have been an increasing development of newer surgical treatment options. Additionally, the outcome parameters for BPH treatments have been somewhat standardized. The purpose of this study is to create an ongoing prospective registry to record demographic data and clinical outcomes after medical therapy or different surgical interventions for BPH. The specific aims of the registry are to analyze demographic patterns and baseline characteristics of men undergoing surgical and medical treatments for BPH, to assess global practice patterns for various surgical and medical treatments of BPH, and to assess key outcomes for uni- and multi-modal treatments of BPH.

The ongoing global registry will provide important baseline data, functional outcomes, and complications following medical and/or surgical intervention for men with symptomatic BPH. The intention of the registry is to provide real world usage data that may be used for future investigations. It will allow providers to identify areas of interest, areas of unusually low usage or areas of unusual preference on a global scale. It will also shed light on global preferences for unimodal or multimodal approaches to treatments.

The registry has been developed using novel database technology, providing an easy-to-use user interface, which enables future creation of patient portals and Electronic Medical Record (EMR) integration.

As this is not an experimental setting, there will be no interventions made on behalf of the registry.

This is a prospective longitudinal ongoing registry. The study will include medical records of all men ≥18 years old who have a primary diagnosis of BPH with Lower Urinary Tract Symptoms (LUTS) that are prescribed BPH medications, or a surgical intervention. Data extraction includes baseline data, peri-operative data, and follow-up data. Baseline data includes validated patient reported outcome tools, including International Prostate Symptom Score (IPSS), Sexual Health Inventory for Men (SHIM), Male Sexual Health Questionnaire - Ejaculatory Dysfunction (MSHQ-EjD), as well as Quality of Life (QoL), maximum flow rate (Qmax), Post-void residual (PVR), Prostate Specific Antigen (PSA), and Testosterone. Complications such as Bleeding, Urinary Tract Infection (UTI), Incontinence, Stricture, Retrograde ejaculation, and Erectile Dysfunction (ED) are also tracked from Baseline through Follow-up.

The registry will run for 3 years with no end point for follow-up. For three years, various research studies will be formulated, and the results will be published. The possibility of extending the study for continued follow-up will be evaluated.

A built-in quality control using data validation during the input process decreases the chance that invalid data will be entered or that datapoints will be omitted. Periodic audits will be performed to verify accuracy of source data by our audit committee based on our audit committee guidelines.

Records and cases of all men with a primary diagnosis of BPH with LUTS that are prescribed BPH medications, or a surgical intervention will be identified and included in the registry. All data is hashed (i.e., protected from decryption) except for a medical record number (MRN), which will be used to add follow-up data to the patient's record. This number is encrypted and linked to the hashed and randomly generated institution code. For security purposes, biographical information is not saved on the registry.

The registry provides secure access to registered users using a web browser. Registrations are site-specific, which means that users can only access the data that is specific to their own site. The registry application and databases are hosted on secure, encrypted servers behind a firewall. They can only be accessed by registered users via a specific port.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of BPH with LUTS with prescribed medical treatment or surgical intervention

Exclusion Criteria:

* Non-symptomatic BPH
* No treatment prescribed for BPH

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years with symptomatic BPH with LUTS who are planned for medical or surgical intervention are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 36 months
  Comparison of mean IPSS score change between baseline and at each follow-up during the course of the study. The scale goes from 0 (Mild) to 35 (Severe).
Quality of Life (QoL) | 36 months
  Comparison of mean QoL score change between baseline and at each follow-up during the course of the study. The scale is a single question which ranges from 0 to 6, with higher numbers indicating a worse quality of life.
Post-Void Residual (PVR) | 36 months
  Comparison of mean PVR change between baseline and at each follow-up during the course of the study.
Complications (including incontinence) | 36 months
  Type and Clavien grade incidences across all surgical interventions.

SECONDARY OUTCOMES:
Prostate Volume (cc) | 36 months
  Comparison of mean Prostate Volume change between baseline and at each follow-up during the course of the study.
Qmax | 36 months
  Comparison of mean Qmax change between baseline and at each follow-up during the course of the study.
Male Sexual Health Questionnaire Ejaculatory Dysfunction (MSHQ-EjD) | 36 months
  Comparison of mean MSHQ-EjD score change between baseline and at each follow-up during the course of the study. The scale ranges from 1 to 15 with a higher score indicating better sexual functioning.
Sexual Health Inventory for Men (SHIM) | 36 months
  Comparison of mean SHIM score change between baseline and at each follow-up during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Desai, MD, Principal Investigator — University of Southern California
Locations (23):
- Keck Medicine of USC, Los Angeles, California, United States
- Canada (2):
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Chile (2):
  - Hospital Dr. Juan Morey La Unión, La Unión
  - Hospital del Trabajador, Santiago
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China
- University of Cyprus, Nicosia, Cyprus
- Shariati Hospital, Tehran, Iran
- University of Basrah, Basra, Iraq
- Italy (2):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Sapienza University of Rome, Division of Urology, Ospedale Sant'Andrea, Rome
- American University of Beirut, Beirut, Lebanon
- Universiti Malaya, Kuala Lumpur, Malaysia
- Kati University Hospital, Kati, Mali
- Centro Medico Nacional Siglo XXI, Mexico City, Mexico
- Nigeria (2):
  - Benue State University Teaching Hospital, Department of Surgery, Makurdi
  - Ahmadu Bello University Teaching Hospital, Zaria
- Pakistan (2):
  - Institute of Kidney Diseases Peshawar, Peshawar
  - Lady Reading Hospital, Peshawar
- Hamad Medical Corporation Qatar, Doha, Qatar
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - Southend University Hospital, Southend-on-Sea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home page — https://www.siu-urology.org/ucare/browse-projects?v=OHtMzjwVVbdmyogNur574NKjMSljFkfy